CLINICAL TRIAL: NCT02396459
Title: Tiratricol Treatment of Children with Monocarboxylate Transporter 8 Deficiency: Triac Trial II
Brief Title: Triac Trial II in MCT8 Deficiency Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rare Thyroid Therapeutics International AB (Industry)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT8-2019-2
Record Dates: First submitted 2015-03-07; First posted 2015-03-24 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Allan-Herndon-Dudley Syndrome
Keywords: Triac; MCT8; MCT8 deficiency; Allan-Herndon-Dudley Syndrome
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome | interventions — 3,3',5-triiodothyroacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MCT8 deficiency patients (Experimental): Triac treatment
  Interventions: Drug: Triac

INTERVENTIONS:
Drug: Triac — Triac, individually titrated dose
  Other Names: Tiratricol; Teatrois

SUMMARY:
This study will investigate the effect of treatment with tiratricol (also called Triac) in young boys (≤30 months) with MCT8 deficiency (also called the Allan-Herndon-Dudley syndrome (AHDS)). The hypothesis tested is that treatment with tiratricol will have a beneficial effect on the hypothyroid state in the brain as well as the hyperthyroid state in peripheral organs and tissues in these patients. Patients will initially be treated for 96 weeks with tiratricol, treatment effect on neurodevelopment impairment caused by hypothyroidism and peripheral thyrotoxicosis will be evaluated after 96 weeks treatment. Patients will be offered to continue on treatment for an additional 2 years.

DETAILED DESCRIPTION:
This therapeutic trial will be conducted in patients with MCT8 deficiency (also called Allan-Herndon-Dudley Syndrome (AHDS)), which is due to mutations in monocarboxylate transporter (MCT)8. MCT8 is a thyroid hormone transporter which is crucial for the transport of thyroid hormone from the blood into different tissues. Defective MCT8 results in a lack of thyroid hormone (hypothyroidism) in tissues that are dependent on MCT8 for thyroid hormone uptake, such as the brain. Hypothyroidism in the brain results in severe intellectual and motor disability. Another important feature of this disease is the high serum T3 concentrations in the blood. This results in hyperthyroidism in tissues that are not dependent on MCT8 for their thyroid hormone supply. As a result, patients with MCT8 deficiency have clinical features of thyrotoxicosis such as low body weight, elevated heart rate and reduced muscle mass.

Preclinical studies have shown that the T3 analogue tiratricol is transported into cells in an MCT8-independent manner. In animal models mimicking MCT8 deficiency, Triac has been shown to normalize brain development if administrated during early postnatal life.

Recently, Triac Trial I (NCT02060474) has shown that tiratricol treatment in patients with MCT8 deficiency improves key clinical and biochemical features caused by the toxic effects of the high T3 concentrations. No drug related serious adverse events have occurred during Triac Trial I.

This study will investigate the effect of treatment with tiratricol in young boys (≤30 months) with MCT8 deficiency (also called the Allan-Herndon-Dudley syndrome (AHDS)). The hypothesis tested is that treatment with tiratricol will have a beneficial effect on the hypothyroid state in the brain as well as the hyperthyroid state in peripheral organs and tissues in these patients. Patients will initially be treated for 96 weeks with tiratricol, treatment effect will be evaluated after 96 weeks. After the 96 week treatment period, patients will enter Part II of the trial, evaluating long-term treatment. Patients will be followed for an additional 2 years and treatment effect will be evaluated after 3 years and 4 years respectively from start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form from the parents or legal guardian.
* Parents stated willingness to comply with all study procedures and availability for the duration of the study.
* The participant should be aged between 0 and 30 months on the day of inclusion.
* The participant should be male and have a pathogenic mutation in the MCT8 gene.

Exclusion Criteria:

* Previous treatment with tiratricol.
* Previous treatment with LT4 and/or PTU and/or other anti-thyroid medication for a period longer than three months. Patients previously treated with LT4 for a shorter period than 3 months may be included in the study (baseline visit) six weeks (or longer) after last dose of LT4 if two consecutive analyses show stable TFT*. Patients treated with PTU and/or other anti-thyroid medication for a shorter period than three months may be included in the study (baseline visit) six weeks (or longer) after last dose.
* Major illness or recent major surgery (within four weeks of baseline visit 1) unrelated to MCT8 deficiency.
* Known allergic reactions to components of the IMP. Patients with galactose intolerance, Lapp lactase deficiency or malabsorption of glucose or galactose (the IMP contains lactose).
* Treatment with another investigational drug or participation in other interventional trial within three months prior to baseline visit 1.

Max Age: 30 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure 88 (GMFM 88) total score | 96 weeks
  To evaluate the effects of tiratricol on neurodevelopment in young MCT8 deficiency patients, measured by the Gross Motor Function Measure (GMFM)-88 assessment. Potential result values range from 0 to 100%, the latter being representative for a 4-year old healthy child. A high score is equivalent to better/more neurodevelopment and is therefore a better outcome than a low score.
Bayley Scales of Infant Development III Gross Motor Skill Domain score | 96 weeks
  To evaluate the effect of tiratricol treatment on neurodevelopment measured by the Bayley Scales of Infant Development (BSID-III) Gross Motor Skill Domain score. Potential total raw scores range from 0-72, and can be age-adjusted before analysis. A high score is equivalent to better/more neurodevelopment and is therefore a better outcome than a low score

SECONDARY OUTCOMES:
GMFM-88 individual item score 10 and 24. | 96 weeks
  GMFM-88 individual item score 10 ("lifts head upright") and item score 24 ("sit on mat"), GMFM Domain B (Sitting) - summary score of all items 18-37 ; Motor milestone responder analysis of Section 2 of the Hammersmith Infant Neurological Examination (HINE).
Bayley Scales of Infant Development III score. | 96 weeks
  To evaluate the effect of tiratricol treatment on neurodevelopment measured by the Bayley Scales of Infant Development (BSID-III). Five subscales of this assessment will be used: Cognitive, Receptive communication, Expressive communication, Fine motor and Gross motor. Potential total raw scores range from 0-91, 0-49, 0-48, 0-66 and 0-72 respectively, and can be age-adjusted before analysis. A high score is equivalent to better/more neurodevelopment and is therefore a better outcome than a low score. This holds true for all subscales.
Serum T3 concentrations | 96 weeks
  Evaluate the effect of tiratricol on clinical and biochemical thyrotoxic features.
Tissue-specific markers of thyroid state: serum sex-hormone binding globulin concentrations for liver | 96 weeks
  Evaluate the effect of tiratricol on clinical and biochemical thyrotoxic features.
Tissue-specific markers of thyroid state: serum creatine kinase concentrations for muscles | 96 weeks
  Evaluate the effect of tiratricol on clinical and biochemical thyrotoxic features.
Tissue-specific markers of thyroid state: serum creatinine concentrations for kidneys | 96 weeks
  Evaluate the effect of tiratricol on clinical and biochemical thyrotoxic features.
Blood pressure | 96 weeks
  Evaluate the effect of tiratricol on clinical and biochemical thyrotoxic features.
Body weight | 96 weeks
  Evaluate the effect of tiratricol on clinical and biochemical thyrotoxic features.

OTHER OUTCOMES:
Patient Quality of Life by Infant Toddler Quality of Life Questionnaire (ITQoL) | 96 weeks
  To evaluate patient´s quality of life (QoL) by Infant Toddler Quality of Life (ITQoL-SF-47) questionnaire. Item responses are scored, summed, and transformed on a scale from 0 (worst health) to 100 (best health). A high score is equivalent to better parent-reported outcomes and is therefore a better outcome than a low score.
Parent Quality of Life by Parenting Stress index (PSI-4 SF) | 96 weeks
  To evaluate parent's quality of life (QoL) by Parenting Stress Index (PSI-4 SF) questionnaire. Results are given as raw scores, percentiles and T scores, where percentiles are the primary interpretive framework. Results from 16th - 84th percentile = Normal range, 85th - 89th Percentile = High range, 90th Percentile or higher = Clinically significant range.
Evaluate the effect of tiratricol treatment on neurological symptoms (Hammersmith Infant Neurological Exam, HINE) | 96 weeks
  Hammersmith Infant Neurological Exam (HINE)
Evaluate the effect of tiratricol treatment on brain function (optional) (EEG) | 96 weeks
  Brain function outcome (optional) evaluated by EEG
Evaluate the effect of tiratricol treatment on brain function (optional) (BERA) | 96 weeks
  Brain function outcome (optional) evaluated by Brainstem Evoked Response Audiogram (BERA)
Evaluate the effect of tiratricol treatment on brain function (optional) (VEP) | 96 weeks
  Brain function/brain imaging outcome (optional) evaluated by Visual Evoked Potentials (VEP)
Evaluate the effect of tiratricol treatment on brain imaging (optional) | 96 weeks
  Brain imaging outcome (optional) evaluated by MRI/MRS - in patients where this examination is scheduled as part of a clinical praxis (at the discretion of the investigator)
Estimate the elimination half-life of tiratricol in young children, reported in hours (optional and provided a medical reason prevails). | 96 weeks
  Measurement of serum T3 concentrations before and 2, 4, 8 and 24 hours after administration of tiratricol as part of pharmacokinetic profile (optional and provided a medical reason prevails)
Estimate the maximum serum concentration of tiratricol in young children, reported in nmol/L (optional and provided a medical reason prevails). | 96 weeks
  Measurement of serum T3 concentrations before and 2, 4, 8 and 24 hours after administration of tiratricol as part of pharmacokinetic profile (optional and provided a medical reason prevails)
Evaluate the occurrence of episodes of tachycardia caused by the thyrotoxicosis. | 96 weeks
  Evaluation of cardiac rhythm and number of episodes of tachycardia with 24 hour Holter ECG.
Evaluate the occurrence of premature atrial complexes (PACs) caused by the thyrotoxicosis. | 96 weeks
  Evaluation of occurrence of PACs with 24 hour Holter ECG.
Evaluate the occurrence of other arrhythmias caused by the thyrotoxicosis. | 96 weeks
  Descriptive evaluation of occurrence of other arrhythmias with 24 hour Holter ECG.
Evaluate the occurrence of structural cardiac anomalies in patients | 96 weeks
  Evaluation of the occurrence of structural cardiac anomalies using routine trans-thoracic cardiac ultrasound.
Number of participants with Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and discontinuations due to Adverse Events (AEs) | 96 weeks
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE is defined as an AE or suspected adverse reaction that at any dose results in any of the following outcomes: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect. Severity was graded as 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). TEAEs are defined as AEs with onset on or after the time of initiation of study drug administration.
Serum free T4 (FT4) concentrations | 96 weeks
  Evaluate the effect of tiratricol on FT4 concentrations to ensure patient safety.
Serum total T4 (T4) concentrations | 96 weeks
  Evaluate the effect of tiratricol on T4 concentrations to ensure patient safety.
Serum tiratricol concentrations | 96 weeks
  Evaluate tiratricol concentrations in serum, as estimated based on measured T3 concentrations in serum.
Serum thyroid stimulating hormone (TSH) concentrations | 96 weeks
  Evaluate the effect of tiratricol on TSH concentrations to ensure patient safety.
Serum reverse T3 (rT3) concentrations | 96 weeks
  Evaluate the effect of tiratricol on rT3 concentrations to ensure patient safety.
Serum Alanine (Amino) Transaminase (ALAT) concentrations | 96 weeks
  Evaluate the effect of tiratricol on ALAT concentrations to ensure patient safety.
Serum Aspartate (Amino) Transaminase (ASAT) concentrations | 96 weeks
  Evaluate the effect of tiratricol on ASAT concentrations to ensure patient safety
Serum gamma-glutamyl transferase (gGT) concentrations | 96 weeks
  Evaluate the effect of tiratricol on gGT concentrations to ensure patient safety.
Serum alkaline phosphatase concentrations | 96 weeks
  Evaluate the effect of tiratricol on alkaline phosphatase concentrations to ensure patient safety.
Serum albumin concentrations | 96 weeks
  Evaluate the effect of tiratricol on albumin concentrations to ensure patient safety.
Serum urea concentrations | 96 weeks
  Evaluate the effect of tiratricol on urea concentrations to ensure patient safety.
Serum sodium concentrations | 96 weeks
  Evaluate the effect of tiratricol on sodium concentrations to ensure patient safety.
Serum potassium concentrations | 96 weeks
  Evaluate the effect of tiratricol on potassium concentrations to ensure patient safety.
White blood cell total and differential count | 96 weeks
  Evaluate the effect of tiratricol on white blood cell total and differential count to ensure patient safety.
Red blood cell count | 96 weeks
  Evaluate the effect of tiratricol on red blood cell count to ensure patient safety.
Platelet count | 96 weeks
  Evaluate the effect of tiratricol on platelet cell count to ensure patient safety.

CONTACTS AND LOCATIONS:
Overall Officials: W.E. Visser, MD, PhD, Principal Investigator — Erasmus Medical Center; Kristina Sjöblom Nygren, MD, Study Director — Rare Thyroid Therapeutics International AB; Stephen LaFranchi_Nicol, Principal Investigator — Oregon Health& Science University (OHSU) Doernbecher Childrens Hospital; Jan Lebl, Principal Investigator — Charles University and Motol University Hospital; Heiko Krude, Principal Investigator — Charité - Universitätsmedizin Berlin Institut fur experimental paediatrische endokrinologie; Andrew Bauer, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (2):
  - Oregon Health & Science University (OHSU) Doernbecher Childrens Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Charles University and Motol University Hospital; The department of peadiatrics of the 2nd faculty of medicine, Prague, Czechia
- Charité - Universitätsmedizin Berlin Institut fur experimental paediatrische endokrinologie, Berlin, Germany
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Because of the rarity of MCT8 deficiency and the small number of patients in this trial, individual patient data beyond what is reported in the upcoming manuscript will not be shared to safeguard patient privacy.